CLINICAL TRIAL: NCT00268814
Title: Phase III Study of Maintenance Treatment for Opiate Dependence With Heroin (Diamorphine) Compared to Methadone
Brief Title: The German Project of Heroin Assisted Treatment of Opiate Dependent Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government); State of Northrhine-Westfalia (Unknown); State of Hessen (Unknown); State of Lower-Saxony (Unknown); City of Hamburg (Other Government); City of Hanover (Other Government); City of Frankfurt (Other Government); City of Bonn (Unknown); City of Cologne (Unknown); City of Munich (Other Government)
Responsible Party: Principal Investigator, PD Dr. Uwe Verthein, Director of Centre for Interdisciplinary Addiction Research, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZIS-HV9-0701
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Heroin; Counseling; Methadone; Case Management; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- MTF, Psycho-education, Heroin (Experimental): Stratum: Methadone treatment failures (MTF) Intervention: Psycho-education and Counselling, Drug: Diacetylmorphine (i.v.)
  Interventions: Drug: Diacetylmorphine; Behavioral: Psycho-education and Counselling
- MTF, Case management, Heroin (Experimental): Stratum: Methadone treatment failures (MTF) Intervention: Case Management and Motivational Interviewing, Drug: Diacetylmorphine (i.v.)
  Interventions: Drug: Diacetylmorphine; Behavioral: Case management and Motivational interviewing
- MTF, Psycho-education, Methadone (Active Comparator): Stratum: Methadone treatment failures (MTF) Intervention: Psycho-education and Counselling, Drug: Methadone (p.o.)
  Interventions: Behavioral: Psycho-education and Counselling; Drug: Methadone
- MTF, Case management, Methadone (Active Comparator): Stratum: Methadone treatment failures (MTF) Intervention: Case Management and Motivational Interviewing, Drug: Methadone (p.o.)
  Interventions: Drug: Methadone; Behavioral: Case management and Motivational interviewing
- NIT, Psycho-education, Heroin (Experimental): Stratum: Not in treatment (NIT) Intervention: Psycho-education and Counselling, Drug: Diacetylmorphine (i.v.)
  Interventions: Drug: Diacetylmorphine; Behavioral: Psycho-education and Counselling
- NIT, Case management, Heroin (Experimental): Stratum: Not in treatment (NIT) Intervention: Case Management and Motivational Interviewing, Drug: Diacetylmorphine (i.v.)
  Interventions: Drug: Diacetylmorphine; Behavioral: Case management and Motivational interviewing
- NIT, Psycho-education, Methadone (Active Comparator): Stratum: Not in treatment (NIT) Intervention: Psycho-education and Counselling, Drug: Methadone (p.o.)
  Interventions: Behavioral: Psycho-education and Counselling; Drug: Methadone
- NIT, Case management, Methadone (Active Comparator): Stratum: Not in treatment (NIT) Intervention: Case Management and Motivational Interviewing, Drug: Methadone (p.o.)
  Interventions: Drug: Methadone; Behavioral: Case management and Motivational interviewing

INTERVENTIONS:
Drug: Diacetylmorphine — Diacetylmorphine (i.v.), daily
  Other Names: Heroin
  Arms: MTF, Case management, Heroin; MTF, Psycho-education, Heroin; NIT, Case management, Heroin; NIT, Psycho-education, Heroin
Behavioral: Psycho-education and Counselling — Psycho-educational group therapy and individual counselling
  Arms: MTF, Psycho-education, Heroin; MTF, Psycho-education, Methadone; NIT, Psycho-education, Heroin; NIT, Psycho-education, Methadone
Drug: Methadone — Methadone (p.o.), daily
  Other Names: racemic d,l-methadone
  Arms: MTF, Case management, Methadone; MTF, Psycho-education, Methadone; NIT, Case management, Methadone; NIT, Psycho-education, Methadone
Behavioral: Case management and Motivational interviewing — Individual Case Management combined with Motivational interviewing
  Arms: MTF, Case management, Heroin; MTF, Case management, Methadone; NIT, Case management, Heroin; NIT, Case management, Methadone

SUMMARY:
The study will test the hypotheses that heroin assisted treatment, compared to methadone maintenance treatment, is more effective with regard to

* the improvement of health,
* reduction of illicit drug consumption,
* decrease of criminal behaviour,
* rise in the accessibility and retainment,
* detachment from a social drug context,
* social stabilisation in the sense of new drug-free contacts, improved vocational circumstances, financial security, stabilisation of the living situation,
* enrollment in subsequent treatment in the case of heroin dependent persons who could not be effectively reached or successfully treated so far, and it will check which is the optimal treatment setting with regard to these aims.

The medication is injectable pure heroin (diacetylmorphine) 3x/d, or d l methadone 1x/d

The study design is multicentre, open, randomised, 4 x 2 stratified. The study duration is 24 months (individual period of investigation), 1. study phase: 12 moths (protocol part B) and 2. study phase: 12 moths (part C). Patients recruited have an opiate dependency according to ICD-10, who are not being treated currently or who are in a methadone maintenance programme with an unsatisfactory course of treatment.

DETAILED DESCRIPTION:
Detailed description of study phase 1 (randomized, controlled part of study) only.

Part B - Study phase 1 B1.1 Clinical hypothesis Compared to maintenance with oral methadone, heroin treatment leads to

* significant improvement of the physical and/or mental state of health,
* greater reduction of illicit drug use and therefore greater detachment from the drug scene,
* significant improvement of the social situation,
* higher retention rate or attachment to treatment, in the case of those heroin dependent persons who could not be effectively reached or could not sufficiently profit from methadone maintenance programmes.

B1.2 Primary outcome criteria

* Improvement of the physical and mental state of health (A) AND
* Reduction of illicit heroin use and non-increase of cocaine use (B). B1.3 Secondary outcome criteria
* Retention rate
* Reduction of benzodiazepine, amphetamine, alcohol and other drug use
* Reduction of scene contacts / of contacts to other drug consumers
* Decrease of delinquent behaviour
* Stabilisation of housing situation
* Establishment of new social contacts
* Improvement of quality of life
* Mortality rate. B2. STUDY DESIGN Phase 1 of the clinical trial consists in a 4 x 2-branched randomised multicentre study. The sample is stratified and consists on the one hand of heroin dependent persons in methadone maintenance treatment that do not sufficiently profit from treatment (MS), and on the other hand of heroin dependent persons who are currently not being treated for their addiction (NE). Patients of both target groups who meet the admission criteria will be randomised to four arms: experimental groups (MS-E-C) and (NE-E-C): heroin treatment with concurrent case management, experimental groups (MS-E-P) and (NE-E-P): heroin treatment with concurrent psychoeducation/drug counseling and control groups (MS-K-C) and (NE-K-C): methadone treatment with concurrent case management, control groups (MS-K-P) and (NE-K-P): methadone treatment with concurrent psychoeducation/drug counseling.

B2.2 Recruitment of patients The period of registration is not part of the individual study period. A screening is carried out at registration concerning certain inclusion criteria. The patients are given the opportunity of a thorough information concerning the conditions and course of the study.

First of all, patients are asked to sign their consent to participate in the study. This is followed by the indication assessment (T-1) by the study physician and the external interview (EuropASI). Certain (particularly medical) characteristics are again examined at the beginning of treatment (T0).

The regionally responsible study physician will decide on the inclusion in the study. His decision needs the confirmation of a regional committee of experts.

B2.3 Randomisation The allocation to treatment places of the experimental or control group is carried out according to a randomisation code. Randomisation is done separately for both groups (MS and NE) based on permuted blocks of fixed size.

After the evaluation of the indication assessment and the first interview (at T-1), patients who have been recruited and who fulfil the inclusion criteria are then asked to give a second consent of participation in the study, and the results of randomisation will be communicated to them.

B2.4 Course of the study, examinations and times of the investigations The first phase of the clinical trial covers a period of 12 months. All questioning is done in a personal interview ("face to face") with the assurance that all information will be confidential.

All patients who take part in the interviews receive an expense allowance of Euro 15.- for each survey.

A hair sample is already taken at the indication examination (T-1). This allows taking a hair sample fit for analysis at the beginning of treatment (T0) from those patients whose hair was too short at T-1. The CIDI will be carried out after one month of treatment in order to minimise initial influences requiring treatment.

In order to determine the use of illicit heroin, which is a main target criterion, five urine controls will be thoroughly examined by GC/MS both in the 6th and the 12th month of treatment.

B3. PATIENTS The adequate treatment of the questions posed by this study requires a number of at least 140 patients in each test group (4 experimental and 4 control groups). Therefore, the sample size for the entire study will be N=1,120.

B3.1 Inclusion criteria

Patients who fulfil following criteria can be included in the study:

* Minimum age 23 years
* Opiate dependence for at least 5 years
* Current main diagnosis of opiate dependency according to the ICD-10 criteria
* Current daily and predominantly intravenous heroin use or continuing heroin use in maintenance treatment
* Symptoms of physical illness indicating a poor state of health according to the OTI health scale; at least 13 current symptoms must be found OR Current mental symptoms or disturbances, i.e. a standardised GSI value of the SCL-90-R of at least 60 points
* No participation in an addiction treatment programme (a.a. maintenance, inpatient or outpatient treatment) at least within the last 6 months, but documented previous experience with drug therapies OR Negative course of maintenance treatment according to the guidelines of the German Medical Council due to (a) continuous additional use of heroin (50% of the urine samples positive within the last 6 months) or cocaine (harmful use of cocaine/crack according to ICD-10) in a documented maintenance period of at least 6 months with a current maintenance dose of at least 60 mg d l methadone (or 30 mg levomethadone) daily
* Residence in the city (or city state) or region for at least 12 months
* Voluntary participation and ability to comply with the treatment conditions
* Written consent to comply with the treatment conditions. B3.2 Exclusion criteria

Persons with at least one of the following criteria cannot be included in the study:

* Persons who are currently in prison or awaiting trial or who can be expected to be taken into custody within the next 3 months
* Persons who had voluntary phases of abstinence of at least 2 months during the last 12 months
* Known epilepsy or generalised convulsions during the last 12 months
* Hypersensitivity to test substances and additives
* Regular intake of MAO inhibitors
* Serious bronchial asthma, COPD, Cor pulmonale
* Serious cardiac arrhythmia
* Prostatic hypertrophy (with urinary retention)
* Urethral stricture
* Life threatening liver disorders (exogenous hepatic coma)
* Serious renal disorders
* Insulin dependent diabetes mellitus
* Diagnosed malignancies during the last 6 months
* Pregnant women or nursing mothers
* Patients unable to comply with the study conditions, i.e. participation in the therapeutic and scientific programmes, due to serious physical or mental illness
* Patients who are currently participating in another clinical study concerned with the evaluation of an addiction treatment programme.

B3.3 Dropping out of treatment

Participation in the study is voluntary i.e. the patient can withdraw his consent to be treated (and to further participation in the study) at any time. Patients having at least one of the following characteristics are removed from treatment:

* Patients suffering from serious somatic complications in connection with heroin or methadone treatment for whom a continuation of treatment would be irresponsible in the opinion of the test study physician and the safety board
* Patients with abnormally changed laboratory values for whom a continuation of treatment would incur great health risks according to the safety board's decision
* Patients who have not turned up at the treatment centre or who have discontinued the study medication for a period of 14 days (or longer) for self-provoked reasons or without giving reasons
* Patients who are taken into custody for one month or longer
* Heroin patients whose treatment must be discontinued for more than 3 months due to hospitalisation or other special treatments
* Patients who, in the opinion of the study physician, cannot or do not want to comply with the conditions of the model project any longer, i.e. participation in the therapeutic and scientific programme
* In case of violence, threat of violence against persons involved in the project or other patients
* In case of drug trafficking on the premises of the model project
* In case of theft, passing on or sale of prescribed substances. B4. TREATMENT B4.1 Treatment setting Patients will be treated in an outpatient clinic. The setting is based on at least weekly contacts to the treating physician. Detailed physical examinations and blood counts (10 ml for each withdrawal) take place at the start of treatment and after 1, 3, 6 and 12 months. There will be weekly urine analyses (qualitative proofs). In addition, a hair sample will be taken from an inconspicuous place at the back of the head at the beginning of treatment (at admission), after 6 months and at the examination after 12 months. Patients under the influence of alcohol, barbiturates or benzodiazepines can be refused their heroin or methadone dose. If excessive alcohol consumption is suspected (smell of alcohol) a breath test is undertaken. If the breath test is above 0.1, heroin or methadone will be refused.

B4.3 Dose regimen Heroin (in combination with methadone) An additional medication of d-1 methadone at night will be offered from the start, i.e. on the second day of treatment at the earliest. The administration of heroin will occur up to 3 times a day during the opening hours of the setting, in the morning, at noon and in the evening. In accordance with the Swiss and Dutch studies, the maximum daily dose of i.v. heroin will be 1,000 mg, the single dose 400 mg. If methadone is claimed at night, it can be taken on the premises during the evening opening hours or taken out as a drinkable, not injectable single dose. The daily maximum dose of additionally prescribed d,l methadone should not exceed 60 mg. Methadone consumption will be controlled by regular urine analyses.

Heroin will be handed out as injectable single doses (in filled syringes) and administered by the patient himself under observation. Patients should stay in the centre for at least 30 minutes after the injection, in order to control for possible unwanted effects.

The different dose regimens (dose regulation at the beginning of treatment or after interruptions starting from different points, fading out in case of (un-)planned treatment conclusions) are based on methadone daily equivalence doses (MTQ). According to the basic rule of the different dose regimens, an individual dose of i.v. heroin for one day, alone or in combination with oral methadone, must not exceed the MTQ of the previous day by more than 50%.

Methadone Oral methadone will be administered once a day. It is taken on the premises under observation as drinkable, not injectable single dose. There is no fixed maximum daily dose; according to experience, dosages between 40 and 160 mg/d of methadone (in individual cases up to 250 mg/d) must be expected. A 1% methadone HCL solution is recommended.

Dose regimen at the conclusion of treatment The conclusion of treatment is done by a step-by-step discontinuation of i.v. heroin or change to oral methadone. The discontinuation of medication (i.v. heroin alone or in combination with methadone) will be done slowly. Preferably, the reduction should not be more than 10%-20% of the MTQ of the previous day. In most cases discontinuation can be completed within 2 weeks. Possible withdrawal symptoms can be treated by concomitant medication.

B5. VARIABLES B5.1 General patient characteristics General and specific sample characteristics such as gender, age, length of opiate dependency, number of previous treatments, current social situation are documented.

B5.2 Medical examination and prescription data, laboratory parameters The daily amounts of heroin or methadone handed out are registered and all further prescriptions are documented. Medical examinations are documented in the CRF.

B5.3 Pharmacokinetics Since pharmacokinetics, the analgetic effects, the tolerance effects and the addiction potential of heroin are well known and new findings are not to be expected within the framework of this study, the study focuses mainly on questions concerning the effects and safety of medication.

B5.4 Efficacy Primary outcome variables Efficacy is investigated with regard to two primary outcome measures - improvement of the state of health (A) and reduction of illicit drug consumption (B). These criteria will be evaluated independently by the statistical comparative analysis; the success of one treatment in comparison to the other treatment is only proven, if both analyses have significant results pointing in the same direction.

State of health (A)

A1. Physical state of health:

Number of symptoms according to the health scale of the Opiate Treatment Index OTI at T 1 and T12.

VA1n = OTI-Health Scale (0 ≤ VA1n ≤ 50).

A2. Mental state of health:

Global Severity Index GSI of the SCL-90-R at T 1 and T12. VA2n = GSI value (0 ≤ VA2n ≤ 4).

The treatment response concerning the improvement of the state of health is given, if one of the two criteria (VA1 or VA2) shows an improvement and the other criteria shows no aggravation. Improvement and aggravation are defined as follows:

* For the physical state of health (VA1): An improvement is indicated by a decrease on the OTI health scale by at least 20% and at least 4 points if T12 is compared with T-1, an aggravation is an increase of at least 20%.
* For the mental state of health (VA2): An improvement is indicated by a decrease of the GSI value by at least 20% if T12 is compared with T-1, an aggravation is an increase of at least 20%.

Illicit drug consumption (B)

B1. Use of illicit heroin:

Number of illicit heroin-positive urine analyses during the 12 months of treatment, i.e. among the last 5 urine samples before T12.

VB1n = number of positive urine samples (0 ≤ VB1 ≤ 5). If the patient has dropped out of treatment, and results at T12 are missing and the LOCF procedure is not possible because of missing urine samples in the 6th month of treatment, but if at least one follow-up has occurred within the ITT method, the patient's self-reported data on use of illicit heroin (physician-CRF) will be used. If these are also missing, self-reported data from the external interview can be used. This will be based on the number of days with illicit heroin consumption during the last 30 days (VB1') before the corresponding time of investigation.

VB1'n = number of illicit heroin consumption days (0 ≤ VB1' ≤ 30).

B2. Cocaine use:

Cocaine concentration of hair based on hair analyses (HAs) at T-1 and T12 within following proof limits:

VB2 n = cocaine concentration (VB2 n ≥ 1 μg/g). If the patient has dropped out of treatment, if results at T12 are missing and the LOCF procedure is not possible because of missing HA at T6, but if at least one follow-up has occurred within the ITT method, the patient's self-reported data on cocaine consumption (physician-CRF) will be used. If these are also missing, self-reported data from the external interview can be used. This will be based on the number of days with cocaine use during the last 30 days (VB2') before the corresponding time of investigation.

VB2'n = number of cocaine consumption days (0 ≤ VB2' ≤ 30). HA does not represent the frequency but the integral intensity within the (past) period of observation assuming an average hair growth of 10 mm per month. The lower limit of proof is assumed to be 1μg/g. An increase of cocaine consumption can be accurately proven, if the value at T12 has increased by 30% in comparison to T-1. (If the hair is too short - less than 1.5 cm - to take a sample at T-1, it will be done at T0.)

Decrease and non-increase of consumption are defined as follows:

* A decrease of illicit heroin use is assumed to be proven, if not more than 2 of the 5 urine samples tested by GC/MS by the 12th month of treatment are positive. If only 4 urine samples are available by the 12th month of treatment, only one urine sample may be positive to illicit heroin. If only 3 urine samples are available, none may be positive to illicit heroin in order to be rated as response. If fewer urine samples are available by the 12th month of treatment, the analyses at the 6th month will be used (LOCF), proceeding according to the same evaluation pattern. Only if no usable urine analyses of the 6th month of treatment exist, the patient's self-report will be used (VB1'). A reduction of illicit heroin consumption of at least 60% between T-1 and T12 in relation to the number of consumption days during the last 30 days is rated as a response.
* The non-increase of cocaine use is proven by the (provable) cocaine concentration in the hair. If a HA cannot be carried out at T12, the hair sample at T6 will be used (LOCF). Only if a usable HA is neither available at T6 (due to a premature discontinuation of treatment), the patient's self report (VB2') will be used. A decrease or no change (with a tolerance of ± 2 days) of the number of consumption days within the last 30 days between T-1 and T12 is rated as a response. I.e. an increase of the number of days with cocaine consumption during the last month of not more than 2 days compared to T-1 is still rated as a response; only an increase at T12 by more than 2 days is rated as non-response.

It has to be assumed that a certain number of patients will prematurely (before initiation of treatment or within the first 3 months) drop-out of treatment (in the case of methadone about 20% up to 40%, in the case of heroin 10%-20%), but that they can be reached again for the examinations and investigations. These patients can be summoned for examination at the fixed times, but 5 urine samples during the last month will not be available from them. These patients without valid data are rated as non-responders in the heroin group and as "worst case" responders in the methadone group. Thus, because a rather high percentage of dropouts in the control group have to be expected, it would be hardly possible to prove the su¬periority of the experimental treatment. In that case, the (negative) result of the study would be caused by problems attributable to the implementation and measuring circumstances of the target criteria so that the evaluation of changes cannot be carried out adequately. Under the specified evaluation strategy, the procedure of measuring the consumption primary outcome measures exclusively by objective methods cannot be maintained.

If 5 urine samples are required within a defined period and 2 at most may be positive, a deviation of this pattern (e.g. urine samples are missing or cannot be used, the patient does not turn up any more) prevents that the primary outcome measures can be reliably investigated and documented. If this happens at T12, a compensation with data at T6 is possible (LOCF). It must be assumed, however, that dropouts occur most often during the first weeks, days or even im¬mediately before the beginning of treatment so that a great number of patients never reaches point T6 for the necessary objective measuring; therefore, it is not realistic to summon dropouts for urine samples 5 times with weekly intervals during the 6th and the 12th month.

An increase of cocaine use is proven by hair analyses (HA). It must be expected also in this case that, for various reasons, a certain number of patients (though much less) will not provide a hair sample at T6 or T12.

Therefore, missing or not useable data concerning the primary outcome measures of illicit heroin use (VB1) and cocaine use (VB2) respectively will be compensated by the patient's report on his consumption during the last 30 days. This procedure is as objective as possible; results are only compensated by subjective data in exceptional cases (dropouts, incorrect or missing data).

The general treatment response is shown by an improvement of the state of health (physical or mental symptoms) and by a decrease of illicit heroin consumption as well as by the non-increase of cocaine consumption between the beginning of treatment and the conclusion of phase 1 of the study.

B5.5 Safety Serious adverse events (SUE), adverse events (UE) and side effects (UAW) must be recorded consistently throughout the study. Side effects will be investigated quantitatively. At each investigation, following effects and side effects related to intoxication will be examined routinely.

The blood controls carried out within the study will be checked for laboratory test abnormalities. Such changes will be documented in the CRF and added to the adverse events (UE) and, if applicable, to the unwanted side effects (UAW).

B6. STATISTICAL ANALYSES B6.1 Safety analysis Under inclusion of all persons who have been randomised, an analysis of emergencies, adverse events (UE) and serious adverse events (SUE) will be carried out. With regard to such events (prevalence, severity classification) potential group differences will be checked for statistical significance.

B6.2 Efficacy analysis The primary outcome analysis will be carried out according to the "intention to treat" principle (ITT), which includes all randomised patients, i.e. all patients who were assigned to one of the treatment groups after twice repeated written consent. With regard to the 4 x 2-branched study design, a 4-factorial logistic regression model will be used. In case of missing information, the "last observation carried forward" method (LOCF) will be applied.

Primary outcome analysis For the experimental and the control groups, this proof of superiority of heroin will be furnished by a 4-factorial logistic regression model; two separated analyses will be calculated for the criterion "improvement of the state of health" (A) and for the criterion "reduction of illicit drug consumption" (B).

An overall success of the study (proof of the superiority of heroin treatment compared to methadone treatment) is assumed if, both for the main target criterion (A) "improvement of the state of health" and the main target criterion (B) "reduction of illicit drug consumption", a superiority of heroin treatment in comparison to methadone treatment can be proven in the respective logistic regression model with an α-error of 5%.

Primary outcome criterion (A) - Improvement of the state of health:

H0A: OR ≤ 1 (Response rate in heroin treatment ≤ Response rate in methadone treatment), H1A: OR > 1 (Response rate in heroin treatment > Response rate in methadone treatment).

The hypothesis is tested one-tailed with a 2.5% alpha error level.

Primary outcome criterion (B) - reduction of illicit drug consumption:

H0B: OR ≥ 1 (Rate of illegal drug use in heroin treatment ≥ in methadone treatment), H1B: OR < 1 (Rate of illegal drug use in heroin treatment < in methadone treatment).

This hypothesis is also tested one-tailed with a 2.5% alpha error level.

Proof of the overall effect of heroin treatment:

The experimental treatment (controlled heroin treatment) will be rated to be successful, if the logistic regression has following results:

* a response rate for the outcome criterion "improvement of the state of health" (A) signifi¬cantly higher in comparison with the control treatment (methadone maintenance) AND
* a response rate for the outcome criterion "reduction of illicit drug consumption" (B) significantly higher in comparison with the control treatment (methadone maintenance).

Secondary outcome analyses The secondary evaluations are carried out according to the scale levels of the variables or of the indices formed (maintenance rate, drug consumption, scene contacts, delinquency, housing situation, social contacts, quality of life, mortality rate), i. e. by bivariate or multivariate analyses.

B6.3 Sample size determination

The calculation of the sample size is based on following efficacy expectation:

• Primary outcome criterion (A) - improvement of the state of health: Efficacy expectation in control groups: ≤ 30% of responders, Efficacy expectation in experimental groups: > 50% of responders.

• Primary outcome criterion (B) - reduction of illicit drug consumption: Efficacy expectation in control groups: ≤ 30% of responders, Efficacy expectation in experimental groups: > 50% of responders. Within the framework of the 4 x 2-branched study design, each primary outcome criterion will be analysed by a 4-factorial logistic regression analysis. With the (conservative) assump¬tion that both target criteria are stochastically independent, a power of 90% for each main out¬come criterion guarantees that a (multiple) total power of 80% is maintained [(1-β)2 ≈ 0.80 for β = 0.10]. Since the total success of the study is only assumed if treatment effects are evident for both primary outcome measures, a correction of type-1-error is not necessary.

A certain number of patients will (prematurely) drop-out of treatment and not be included in the evaluation by LOCF, because they cannot be reached any more for examinations and interviews. These are patients who dropped out prior to T6 or have not started treatment or refused their consent to the investigation of the two primary outcome variables. According to the conservative evaluation strategy, these patients must be treated as "worst cases". Therefore, the size of the assumed effect decreases in relation to the percentage of these "not reached" patients in the heroin and methadone group. Realistic estimations of these percentages are 10% drop-outs in the methadone group and 5% in the heroin group. According to these expected percentages, the estimated effect size on which the calculation of the sample size is based, is reduced from 0.3 vs. 0.5 to 0.370 vs. 0.475.

Based on this assumption, a multiple total power of 80% requires a number of cases of at least N=482 test persons for each sample group (based on Chi2-test for odds ratio, sample size approximation according to Nam 1992). Related to the individual strata, this means at least four heroin and four methadone strata with at least 121 patients each are necessary to prove the expected effect with a statistical power of 80%. For practical reasons (adequate distribution to the study cen¬tres, increased measuring precision), this number is rounded up to N=140 resulting in eight strata with a total number of N=1,120 patients.

Under the described conditions, this sample size guarantees that in both tests a significant difference between methadone and heroin treatment can be proven with a statistical total power of at least 80%.

B6.4 Missing data If data of the 12-months examination are missing and concern the primary outcome criteria and cannot be replaced by the LOCF method, a non-fulfillment of the criterion must be assumed, which will be interpreted as "worst case" in the individual case.

B6.5 Drop-outs Patients dropping out of treatment will continue to be included in the investigations and evaluations (ITT-analysis). According to the LOCF method, the latest information of each patient will be used for the analysis if a patient cannot be interviewed at the conclusion of the study. As far as the primary outcome criterion of illicit heroin consumption is concerned, the 12-month information can only be completed by the investigation at T6, because only the five urine samples in the 6th month of treatment can be tested for illicit heroin by GC/MS. Similarly, a missing hair analysis for cocaine consumption at T12 can only be completed by a hair sample precautiously taken at T6. If no objective measure results of the primary outcome measures illicit heroin and cocaine consumption are available, the patient's self-report will be included in the analysis.

Patients who did not participate in any further investigation after the inclusion in the study are rated as "worst case", i.e. not reached patients of the methadone group are rated as success (responders) and not reached patients of the heroin group as failures (non-responders). Patients who died in the first phase of the study are rated (in the experimental and the control group) as non-responders. Patients, who withdraw their consent after randomisation and do not initiate the study treatment, are excluded from the ITT-analysis.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 23 years
* Opiate dependency for at least 5 years
* Current main diagnosis of opiate dependency according to the ICD-10 criteria
* Current daily and predominantly intravenous heroin consumption or continuing heroin consumption in maintenance treatment
* Symptoms of physical illness indicating a poor state of health according to the OTI health scale; at least 13 current symptoms must be found OR Current mental symptoms or disturbances, i.e. a standardised GSI value of the SCL-90-R (Franke 1995) of at least 60 points
* No participation in an addiction treatment programme (a.a. maintenance, inpatient or outpatient treatment) at least within the last 6 months, but documented previous experience with drug therapies OR Negative course of maintenance treatment according to the guidelines of the German Medi¬cal Council (Bundesärztekam¬mer 1997) due to (a) continuous additional consumption of heroin (50% of the urine samples positive within the last 6 months) or cocaine (harmful use of cocaine/crack according to ICD-10) in a documented maintenance period of at least 6 months with a current maintenance dose of at least 60 mg d l methadone (or 30 mg levo¬methadone) daily
* Residence or registration in the city (or city state) or region that conducts the heroin treat¬ment for at least 12 months
* Voluntary participation and ability to comply with the treatment conditions (willingness to change treatment location; compliance; treatment control/documentation; evalua¬tion)
* Written consent to comply with the treatment conditions.

Exclusion Criteria:

* Persons who are currently in prison or awaiting trial or who can be expected to be taken into custody within the next 3 months
* Persons who had voluntary phases of abstinence of at least 2 months during the last 12 months
* Known epilepsy or generalised convulsions during the last 12 months
* Hypersensitivity to test substances and additives
* Regular intake of MAO inhibitors
* Serious bronchial asthma, COPD, Cor pulmonale
* Serious cardiac arrhythmia
* Prostatic hypertrophy (with urinary retention)
* Urethral stricture
* Life threatening liver disorders (exogenous hepatic coma)
* Serious renal disorders
* Insulin dependent diabetes mellitus
* Diagnosed malignancies during the last 6 months
* Pregnant women or nursing mothers
* Patients, who, according to the study physician's judgement, are not able to comply with the conditions of the model project, i.e. participation in the therapeutic and scientific pro¬grammes, due to serious physical or mental illness
* Patients who are currently participating in another clinical study concerned with the evalua¬tion of an addiction treatment programme.

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2002-03; Primary Completion 2003-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
(A) Improvement of physical or mental state of health, | 12 months
(B) Reduction of consumption of street heroin and no increase of cocaine use. | 12 months

SECONDARY OUTCOMES:
Retention rate | 12 months
Reduction of consumption of, benzodiazepines, amphetamine, alcohol and other substances | 12 months
Detachment from the drug scene | 12 months
Decrease of criminal behaviour | 12 months
Stabilisation of the living situation | 12 months
Establishment of new social contacts | 12 months
Improvement of quality of life | 12 months
Mortality rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Naber, MD, Principal Investigator — University of Hamburg-Eppendorf; Christian Haasen, MD, Study Director — University of Hamburg-Eppendorf
Locations (7):
- Germany (7):
  - AWO Ambulanz, Karlsruhe, Baden-Wuertenberg
  - Heroinambulanz, Munich, Bavaria
  - Pro Vivere Drogenambulanz, Hamburg, Hamburg
  - Studienambulanz, Frankfurt am Main, Hesse
  - Drogenambulanz Hannover, Hanover, Lower-Syxony
  - Heroinambulanz Bonn, Bonn, Northrhine-Westfalia
  - Heroinambulanz Koeln, Cologne, Northrhine-Westfalia

REFERENCES:
- See also: Webpage with information on the trial — http://www.heroinstudie.de